CLINICAL TRIAL: NCT04970862
Title: Evaluation of the Effect of Revision Surgery of Lumbar Adjacent Segment Degeneration
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020288
Record Dates: First submitted 2021-07-02; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Adjacent Segment Disease; Adjacent Segment Degeneration
Keywords: Adjacent Segment Degeneration; reversion surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: reversion surgery — reversion surgery

SUMMARY:
The purpose of this study was to investigate postoperative imaging changes and clinical symptom improvement in patients undergoing revision surgery for adjacent segment degeneration.

ELIGIBILITY:
Inclusion Criteria:

* For patients undergoing revision surgery in adjacent segments due to S-ASD, the revision surgery is at least half a year from the first operation;
* X-ray, CT and MRI examination data of the anterior and lateral extension of the lumbar spine were available within 1 month before surgery and at the last follow-up;
* Follow-up for at least 2 years after revision;

Exclusion Criteria:

* Patients with history of congenital spinal deformity, spinal tumor, spinal tuberculosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2010 to June 2018, patients with lumbar spine disease hospitalized in orthopedics were screened out to meet the criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) scores of low back pain and leg pain | 2 years after revision surgery
  Visual Analog Scale (VAS) scores of low back pain and leg pain
Japanese Orthopedic Association (JOA) score | 2 years after revision surgery
  Japanese Orthopedic Association (JOA) score
Oswestry Disability Index (ODI) | 2 years after revision surgery
  Oswestry Disability Index (ODI)

CONTACTS AND LOCATIONS:
Overall Officials: Weishi Li, M.D., Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No